CLINICAL TRIAL: NCT02311491
Title: Nano-Crystalline Ceramic Coating for the Reduction of Sliding Resistance of Orthodontic Archwires
Brief Title: Nano-Crystalline Ceramic Coating of Orthodontic Archwires
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding terminated
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: N2 Biomedical LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-0924
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Malocclusion
Keywords: nano crystalline; archwire
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ceramic Coated Orthodontic Archwire (Experimental): Ceramic coated orthodontic archwires will be evaluated in a limited clinical study at the university of North Carolina to test their efficacy in early and intermediate stages of tooth straightening in orthodontic patients.
  Interventions: Device: Ceramic coated orthodontic archwire
- Control (No Intervention): The patients will receive the ordinary archwires. There is no intervention to the standard treatment.

INTERVENTIONS:
Device: Ceramic coated orthodontic archwire — Hard ceramic coatings will reduce the sliding resistance of archwires in their brackets during orthodontic treatment procedures. The new coated archwire is expected to reduce treatment time.
  Arms: Ceramic Coated Orthodontic Archwire

SUMMARY:
Purpose: The project aims to assess if hard ceramic coatings on orthodontic archwires will reduce the sliding resistance of archwires in the brackets during orthodontic treatment procedures.

Participants: Up to 80 subjects will be recruited for this study. Subjects between 10 years of age and 45 years old will be otherwise healthy subjects previously diagnosed with malocclusion.

Procedures (methods): Each subject will receive an experimental (coated) or a regular (uncoated control) orthodontic archwire (AW) for a 3-month treatment. The 3D digital images of each subject's dentition will be recorded three times at 0-, 6- and 12-week visits. The AW will be removed and retrieved after the 3-month trial.

DETAILED DESCRIPTION:
In this trial, nano-crystalline ceramics will be applied to the surface of orthodontic archwires using ion beam assisted deposition to reduce sliding resistance. Excessive sliding resistance works against tooth motion as the bracket slides along the wire into a new position. These ceramic coatings will produce more predictable outcomes, requiring less force and shorter treatment time. A limited clinical trial will be conducted to demonstrate these effects.

The aim of this project is to assess the clinical efficacy of the new archwires in Stage 1 (leveling and aligning) and Stage 2 (space closure) of orthodontic treatment using a twin bracket. The working hypothesis is that reduction of sliding resistance in bracket-wire interfaces will allow effective tooth movement in leveling, aligning, and sliding, while minimizing unwanted tooth movement such as lateral (mesio-distal direction) movement due to friction. This will be tested in a total of 80 patients who are undergoing active treatment in the University of North Carolina (UNC) orthodontic graduate clinic. These patients will be comprised of a treatment group (coated) and a control group (uncoated) of 20 each in Stage 1 and Stage 2 treatment.

A successful program will demonstrate a clinically significant increase in the amount and rate-of-change of tooth movement in leveling, aligning, and sliding teeth.

ELIGIBILITY:
Inclusion Criteria:

In the initial or second stage of active treatment at the University of North Carolina graduate orthodontic clinic

Specific inclusion criteria for 1st order tooth movement:

1. Non-extraction treatment in mandible
2. Mandibular Little Index greater than or equal to 5 mm
3. Presence of all permanent anterior teeth
4. Age 10-45 years
5. Consent to participate in the study

Specific inclusion criteria for 2nd order tooth movement:

1. Space closure treatment need greater than or equal to 3 mm (extraction and/or non-extraction patients)
2. Space closure being carried out via sliding mechanics using power chains, spring coils, or interarch elastics
3. Age 10-45 years
4. Consent to participate in the study

Exclusion Criteria:

Specific exclusion criteria for 1st order tooth movement:

1. Systemic diseases such as diabetes, hypertension, temporomandibular disorders (TMD), craniofacial syndrome, etc.
2. Subjects who have incisor mandibular plane angle (IMPA) greater than or equal to 100 degrees
3. Anterior tooth completely blocked from the arch form
4. Periodontal pocketing of any lower anterior teeth greater than 4 mm

Specific exclusion criteria for 2nd order tooth movement:

1. Systemic diseases such as diabetes, hypertension, TMD, craniofacial syndrome, etc.
2. Space closure being carried out via closing loops
3. Periodontal pocketing greater than 4 mm

Ages: 10 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Effective tooth movement in translation | 12 weeks
  Clinical linear measurements (mm) in x-, y-, and z-translation at three time points (0-, 6-, and 12-weeks). A repeated measurement ANOVA model for the continuous clinical outcomes will be considered to test the proposed hypotheses.
Effective tooth movement in rotation | 12 weeks
  Clinical angular measurements (degree) in x-, y-, and z-rotation at three time points (0-, 6-, and 12-weeks). A repeated measurement ANOVA model for the continuous clinical outcomes will be considered to test the proposed hypotheses.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Chang Ko, DDS, PhD, Principal Investigator — UNC-CH